CLINICAL TRIAL: NCT05519410
Title: A Prospective, Two-arm, Randomized，Phase II Clinical Study of Sintilimab Combined With Lenvatinib Versus Hepatic Artery Infusion Chemotherapy for Perioperative Treatment of Resectable Primary Hepatocellular Carcinoma With a High Risk of Recurrence.
Brief Title: Sintilimab Combined With Lenvatinib Versus HAIC for Perioperative Treatment of Resectable Primary Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2022-08-23; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Resectable Hepatocellular Carcinoma
MeSH Terms: interventions — sintilimab; lenvatinib

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab Combined With Lenvatinib (Experimental): Pre-operation: 2-3 cycles;
  Interventions: Drug: Sintilimab and Lenvatinib
- HAIC (Active Comparator): Pre-operation: HAIC-FOLFOX 2-3 cycles;
  Interventions: Drug: HAIC-FOLFOX

INTERVENTIONS:
Drug: Sintilimab and Lenvatinib — Tislelizumab, 200mg, ivd,q3w; Lenvatinib,8mg/kg,po,qd.
  Arms: Sintilimab Combined With Lenvatinib
Drug: HAIC-FOLFOX — hepatic artery infusion Oxa 85 mg/m2, CF 400 mg/m2, 5-Fu 400 mg/m2, 5-Fu 2400mg/m2 infusion 48h.
  Arms: HAIC

SUMMARY:
This is a prospective, Two-arm, randomized，phase II clinical study of Sintilimab Combined With Lenvatinib Versus HAIC for perioperative treatment of resectable primary hepatocellular carcinoma with a high risk of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients volunteered to participate in this study and signed informed consent;
* Age 18-75, male or female;
* ECOG PS score 0-1;
* Child-pugh liver function grading: Grade A
* The clinical diagnosis conforms to primary hepatocellular carcinoma (HCC) and the lesion conforms to the indications for resectable operation in the Guidelines for diagnosis and Treatment of HCC (2019) edition;
* According to the preoperative evaluation of the researcher, the patient had a high risk of recurrence and met at least one of the risk factors:

  * b: 2-3 tumors with the maximum diameter ≤3cm; IIa: tumor 2-3,biggest > 3 cm in diameter
* According to RECIST 1.1 standard, patients have at least one measurable lesion (CT/MRI scan long diameter ≥10mm or CT/MRI scan short diameter ≥15mm for lymph node lesions, and the lesion has not received radiotherapy, freezing or other local treatments);
* Expected survival ≥ 6 months;
* The function of vital organs meets the following requirements (excluding the use of any blood component and cell growth factor within 14 days) ;
* Blood routine:

Neutrophils ≥1.5×109//L Platelet count ≥100×109/L Hemoglobin ≥90g/L;

-Liver and kidney function: Serum creatinine (SCr) ≤ 1.5 times upper limit of normal value (ULN) or creatinine clearance ≥50 ml/min (Cockcroft-Gault formula); Total bilirubin (TBIL)≤ 1.5 times the upper limit of normal value (ULN); AST or ALT levels ≤ 2.5 times the upper limit of normal value (ULN); Urine protein <2+;If urinary protein ≥2+,24-hour quantitative urine protein must be ≤1g;

* Normal coagulation function, no active bleeding and thrombotic disease A. International standardized ratio INR≤1.5×ULN; B. Partial thromboplastin time APTT≤1.5×ULN; C. Prothrombin time PT≤1.5ULN;
* Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during and within six months of the end of medication; Patients with negative serum or urine pregnancy tests within 7 days prior to study inclusion and who must be non-lactating, and males should agree to use contraceptives during the study period and for 6 months after the end of the study period;
* Subjects have good compliance and cooperate with the follow-up.

Exclusion Criteria:

* Have received radiotherapy, chemotherapy, concurrent chemoradiotherapy or other targeted therapies before;
* Known hepatobiliary cell carcinoma, sarcomatoid hepatocellular carcinoma, mixed cell carcinoma and fibre-lamellar cell carcinoma; Active malignancies other than HCC within 5 years or concurrently;
* Having hypertension that cannot be well controlled by antihypertensive drug therapy (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);Previous history of hypertension crisis or hypertensive encephalopathy;
* Subject has previous or concurrent malignancies (except cured basal cell carcinoma of skin and carcinoma in situ of the cervix);
* Previous treatment with Tislelizumab or other PD-1/PD-L1 treatment could not be enrolled; Subjects are known to have prior allergies to macromolecular protein reparations or to any Tislelizumab or Lenvatinib excipients;
* Subject has any active autoimmune disease or history of autoimmune disease (such as, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism; Subjects with vitiligo or childhood asthma have been completely relieved and may be included as adults without any intervention; Asthma requiring medical intervention with bronchodilators will not be included);
* Subjects are receiving immunosuppressive, or systemic, or absorbable local hormone therapy for immunosuppression purposes (>10mg/ day prednisone or other therapeutic hormones) and continue to receive such therapy within 2 weeks prior to enrollment;
* Ascites or pleural effusion with clinical symptoms require therapeutic puncture or drainage;
* Clinical symptoms or diseases of the heart that are not well controlled, such as:

NYHA2 or above heart failure Unstable angina pectoris Myocardial infarction occurred within 1 year

* Patients with clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention;
* The patient currently (within 3 months) has gastrointestinal diseases such as esophageal varices, active gastric and duodenal ulcers, ulcerative colitis, portal hypertension, or active bleeding in unresected tumors, or other conditions determined by the researchers that may cause gastrointestinal bleeding or perforation;
* Past or present severe bleeding (>30 ml bleeding within 3 months), hemoptysis (>5 ml fresh blood within 4 weeks) or thromboembolic events (including stroke events and/or tia) within 12 months;
* Subject has active infection or unexplained fever of >38.5 degrees during screening and before first administration (subject's fever due to tumor can be enrolled according to the investigator's judgment);
* Patients with past or present objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radioactive pneumonia, drug related pneumonia, severe impairment of lung function, etc.;
* Subjects with congenital or acquired immune deficiency, such as HIV infection, or active hepatitis (transaminase does not meet the inclusion criteria, hepatitis B reference: HBV DNA≥1000/ml; Hepatitis C reference: HCV RNA≥103/ml);Chronic hepatitis B virus carriers, HBV DNA < 1000 IU/ml, must receive antiviral treatment at the same time during the test can be enrolled;
* Live vaccine is administered less than 4 weeks before or possibly during the study period;
* The subject has a known history of psychotropic substance abuse, alcohol abuse or drug abuse;
* The subject cannot or does not agree to bear the cost of the self-funded portion of the examination and treatment, except for the clinical study drug, combined chemotherapy and SAE related to the clinical study drug combined chemotherapy; Researchers think that should be left out in this study, the researchers determine, for example, the subjects have other factors that may result in this study were forced to midway termination, such as, other serious disease (including mental illness) need to merge treatment, there are serious abnormal laboratory examination, accompanied by factors such as family or society, will affect the safety of the subjects, or information and the collection of the sample.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-23 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
1-year DFS% | 12month
  1-year disease-free survival rate

SECONDARY OUTCOMES:
ORR | 3 months
  objective response rate
Percentage of MVI | 4 months
  Microvascular invasion
Percentage of pCR | 4 months
  pathological complete response
2-year DFS% | 24 months
  2-year disease-free survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China